CLINICAL TRIAL: NCT04125368
Title: A Feasibility Study of Integrating Maternal Nutrition Interventions Into Antenatal Care Services in Ethiopia: A Cluster-Randomized Evaluation
Brief Title: A Feasibility Study of Integrating Maternal Nutrition Interventions Into Antenatal Care Services in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Addis Continental Institute of Public Health (Other); FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHND-19-0948
Record Dates: First submitted 2019-10-08; First posted 2019-10-14 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Maternal Dietary Diversity; Iron-Folic Acid Supplementation; Early Initiation of Breastfeeding
Keywords: Maternal Nutrition; Antenatal Care; Ethiopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A&T intervention areas: intensified maternal nutrition behavior change interventions during antenatal care delivered through government health facilities and in the community
  Interventions: Behavioral: Health Facility Interventions; Behavioral: Community Interventions; Behavioral: Health System Interventions
- Control (No Intervention): Comparison areas: standard antenatal care services delivered at government health facilities and in the community

INTERVENTIONS:
Behavioral: Health Facility Interventions — 1. Intensified counselling on dietary diversity and increased meal frequency during pregnancy.
  2. Strengthened government distribution of IFA supplies with counseling about its importance, managing side effects, and reminder about subsequent supplies.
  3. Weight-gain monitoring with messaging to mothers about healthy diet and adequate rest; excess weight gain as a danger sign.
  4. Intensified counseling on importance, benefits, and how-tos of early initiation of breastfeeding and exclusive breastfeeding.
  Arms: Intervention
Behavioral: Community Interventions — 1. Home visits to pregnant women by HEWs to discuss maternal nutrition (dietary diversity, adequate food intake, IFA supplementation, and weight gain), early breastfeeding practices, provide ANC and Pregnant Women Conference referrals, and engage husbands.
  2. HEWs use A&T intervention tools (e.g. posters and maternal nutrition follow-up card) at Pregnant Women Conferences/ Mother Support Groups to reinforce maternal nutrition messages, encourage ANC attendance, distribute IFA tablets, measure and track weight gain, promote early breastfeeding practices, and encourage husband participation.
  3. HEWs and community volunteers (Women's Development Army (WDA), imams, etc.) deliver maternal nutrition messages and encourage ANC visits at kebele and community meetings.
  Arms: Intervention
Behavioral: Health System Interventions — 1. Trainings on the maternal nutrition interventions for health center heads, nurse-midwives, HEWs, community volunteers (WDA, imams, etc.), woreda health officers, and other key actors.
  2. Supportive supervision of maternal nutrition activities conducted by woreda nutrition officers, woreda health officers, TDA or A&T.
  Arms: Intervention

SUMMARY:
Alive & Thrive (A&T) is an initiative that supports the scaling up of nutrition interventions to save lives, prevent illnesses, and contribute to healthy growth and development through improved maternal nutrition, breastfeeding and complementary feeding practices. In Ethiopia, A&T integrated a package of maternal nutrition interventions into existing antenatal care (ANC) services delivered through government health facilities (counselling on diet quality during pregnancy, distribution and promotion of iron-folic acid (IFA) supplementation, weight gain monitoring, counselling on early breastfeeding practices, and systems strengthening through training and supportive supervision) and community platforms (home visits, Pregnant Women Conferences/Mother Support groups, and community gatherings). The evaluation used a two-arm cluster-randomized, non-masked trial design, consisting of two cross-sectional surveys in 2019 and 2021.

DETAILED DESCRIPTION:
There is wide recognition of the importance of integrating maternal nutrition interventions in ANC to improve maternal and child health. In 2016, World Health Organization ANC guidelines were updated to place a high priority on nutrition interventions during pregnancy to improve perinatal outcomes and women's experience of care.

In Ethiopia, the government has adopted a package of maternal nutrition interventions into national guidelines (see Ethiopia's Federal Ministry of Health National Guideline on Adolescent, Maternal, Infant and Young Child Nutrition). Despite these efforts, the coverage and quality of maternal nutrition interventions remains low.

A&T Ethiopia integrated a package of maternal nutrition interventions into existing ANC services delivered through government health facilities (counselling on diet quality during pregnancy, distribution and promotion of IFA supplementation, weight gain monitoring, counselling on early breastfeeding practices, and systems strengthening through training and supportive supervision) and community platforms (home visits, Pregnant Women Conferences/Mother Support groups, and community gatherings) that align with the latest global evidence. IFPRI tested the feasibility of the behavior-change interventions and examined their impacts on pregnant women's health and nutrition practices and breastfeeding practices of recently delivered women, compared with standard antenatal care services provided in control areas.

The evaluation used a two-arm cluster-randomized, non-masked trial design, consisting of two cross-sectional surveys of pregnant and recently delivered women who attended government ANC services. The unit of randomization is the health center and associated health posts in the catchment area. 18 health centers and 2 hospitals in SNNPR and 10 health centers in Somali were randomly assigned to intervention/control. The baseline survey was conducted in October-November 2019, and the endline survey took place in July-September 2021. In 2020, program activities were interrupted between April and July 2020 due to the COVID-19 pandemic. The endline survey was postponed to July-September 2021 to maximize implementation duration.

The overall study objective was to determine the feasibility and impact of integrating locally relevant maternal nutrition interventions into existing ANC services on diet quality and utilization of nutrition interventions during pregnancy.

Research questions include:

1. What are the program impacts on maternal practices: (1) consumption of diversified foods during pregnancy; (2) consumption of IFA supplements during pregnancy; and (3) early breastfeeding practices?
2. Can the coverage and utilization of key maternal nutrition interventions during ANC be improved through system strengthening approaches?
3. What factors influenced the integration and strengthening of maternal nutrition interventions into the government ANC service delivery platform?

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant or recently delivered with a child 0-5.9 months of age
* Attended at least 1 ANC visit at a government health center or health post
* Resides in the same kebeles as the government health center catchment area
* Given informed consent
* Service providers and health facilities in the catchment areas

Exclusion Criteria:

* Age <15 years or >49 years

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 4256 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-04 (Actual)

PRIMARY OUTCOMES:
Dietary diversity during pregnancy | Approximately 2 years after baseline in a cross-sectional endline survey
  Mean number of food groups consumed by pregnant women on the day preceding the interview.
Minimum dietary diversity during pregnancy | Approximately 2 years after baseline in a cross-sectional endline survey
  Proportion of pregnant women who consumed 5 or more food groups on the day preceding the interview.
Consumption of iron-folic acid tablets during pregnancy | Approximately 2 years after baseline in a cross-sectional endline survey
  Mean number of IFA tablets consumed during last pregnancy by recently delivered women with a child 0-5.9 months of age.
Consumption of 90+ iron-folic acid tablets during pregnancy | Approximately 2 years after baseline in a cross-sectional endline survey
  Proportion of women who consumed 90+ IFA supplements during pregnancy by recently delivered women with a child 0-5.9 months of age.

SECONDARY OUTCOMES:
Early initiation of breastfeeding | Approximately 2 years after baseline in a cross-sectional endline survey
  Proportion of children aged 0-5.9 months who were breastfed within 1 hour of birth.
Use of ANC services during pregnancy | Approximately 2 years after baseline in a cross-sectional endline survey
  Total number of ANC visits and month of first ANC visit during last pregnancy reported by recently delivered women with a child age 0-5.9 months.
Exposure to maternal nutrition interventions from ANC | Approximately 2 years after baseline in a cross-sectional endline survey
  Proportion of recently delivered women with children <6 months of age exposed to maternal nutrition interventions from ANC and other sources.
Women's knowledge of maternal nutrition and breastfeeding | Approximately 2 years after baseline in a cross-sectional endline survey
  Proportion of recently delivered women with children <6 months of age with correct knowledge of maternal nutrition and appropriate breastfeeding practices based on survey responses.
Health worker knowledge of IFA supplementation, dietary diversity, weight gain during pregnancy, and early initiation of and exclusive breastfeeding. | Approximately 2 years after baseline in a cross-sectional endline survey
  Proportion of nurse-midwives and health extension workers with correct knowledge of IFA supplementation, dietary diversity, weight gain during pregnancy and appropriate breastfeeding practices based on survey responses.
Availability of ANC service supports | Approximately 2 years after baseline in a cross-sectional endline survey
  Proportion of health facilities with service supports (IFA supplies, records/registers and regular review of nutrition intervention coverage and IFA supply data, weight measurement equipment, counseling materials, and training and supervision for health workers) based on enumerator observation.

CONTACTS AND LOCATIONS:
Locations (1):
- International Food Policy Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
In compliance with donor open access policy requirements, fully anonymized datasets will be made publicly available one year after the end of the project. Metadata and other documentation of data collection procedures (such as the codebook, data collection instruments and interviewer guides/protocols) will also be made publicly available.
Supporting Information: Study Protocol
Time Frame: Fully anonymized datasets will be made publicly available one year after the end of the project.

DOCUMENTS (3):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04125368/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT04125368/SAP_001.pdf
  • Informed Consent Form (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04125368/ICF_002.pdf